CLINICAL TRIAL: NCT03479723
Title: Identification of Predictors for Coronary Plaque Erosion in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine; Director, Cardiology Laboratory for Integrative Physiology & Imaging, Massachusetts General Hospital
Other Study IDs: 2017P000329
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to perform pooled analysis with data collected from 5 previously published studies and 8 unpublished datasets collected from international sites. The main goal of this study is to identify the predictors of plaque erosion.

DETAILED DESCRIPTION:
Plaque erosion is reported to be responsible for about one third of patients with acute coronary syndrome (ACS). In the EROSION study, we reported that antithrombotic therapy without stenting achieved a reduction in thrombus volume greater than 50% in over 70% of patients diagnosed with ACS caused by plaque erosion. This result suggests that the conservative approach of anti-thrombotic therapy without stenting may be an option for patients diagnosed with ACS caused by plaque erosion, which may be the paradigm shift in treatment of ACS patients. However, at present, the only way to make an in vivo diagnosis of plaque erosion is intra-coronary optical coherence tomography (OCT). If we can identify clinical factors associated with plaque erosion, we may be able to narrow down a sub-population of patients with a higher likelihood of plaque erosion. This group of patients may be stabilized with pharmacologic therapy and avoid invasive procedures, thereby preventing related complications and reducing health care burden. However, specific demographic characteristics of the ACS patients with plaque erosion are not known. Our group has the world's largest dataset of patients with plaque erosion and several published reports on plaque erosion. However, the study population of each study is still small and unbalanced to identify the demographic characteristics associated with plaque erosion. Therefore, we propose to pool data from a large number of institutions around the world. This will provide an opportunity to identify factors associated with plaque erosion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ACS upon admission to hospital, including patients with ST-elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), and unstable angina pectoris (UAP).
2. Intra-vascular OCT imaging of culprit vessel.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of ACS confirmed by OCT imaging of the culprit lesion.
Sampling Method: Probability Sample
Enrollment: 1793 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Cardiac death | 3-year

SECONDARY OUTCOMES:
all cause death | 3-year
myocardial infarction | 3-year
stent thrombosis | 3-year
  stent thrombosis was defined according to the Academic Research Consortium criteria
any target lesion revascularization | 3-year
  Any revascularization due to thrombosis or restenosis of the target lesion
clinically driven target lesion revascularization | 3-year
  target lesion revascularization performed because of ischemic symptoms, electrocardiographic changes at rest or positive stress test relists
target-vessel revascularization | 3-year
  Revascularization of any segment of the coronary artery containing the target lesion
any repeat revascularization | 3-year
stroke | 3-year
device-oriented composite (cardiac death, target vessel MI, and TLR) | 3-year
bleeding complication | 3-year
  Gusto and BARC definition
patients-oriented composite (all cause death, MI, any repeat coronary revascularization) | 3-year
target vessel failure (TVF; cardiac death, MI, or ischemia-driven TVR) | 3-year
major adverse cardiac events (MACEs: cardiac death, MI, or ischemia-driven TLR) | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Suzuki K, Niida T, Yuki H, Kinoshita D, Fujimoto D, Lee H, McNulty I, Takano M, Nakamura S, Kakuta T, Mizuno K, Jang IK. Coronary Plaque Characteristics and Underlying Mechanism of Acute Coronary Syndromes in Different Age Groups of Patients With Diabetes. J Am Heart Assoc. 2023 Dec 5;12(23):e031474. doi: 10.1161/JAHA.123.031474. Epub 2023 Nov 28. PMID 38014673
- [Derived] Seegers LM, Yeh DD, Wood MJ, Yonetsu T, Minami Y, Araki M, Nakajima A, Yuki H, Ako J, Soeda T, Kurihara O, Higuma T, Kimura S, Adriaenssens T, Nef HM, Lee H, McNulty I, Sugiyama T, Kakuta T, Jang IK. Cardiovascular Risk Factors and Culprit Plaque Characteristics in Women With Acute Coronary Syndromes. Am J Cardiol. 2023 Nov 15;207:13-20. doi: 10.1016/j.amjcard.2023.08.152. Epub 2023 Sep 16. PMID 37722196
- [Derived] Yuki H, Kinoshita D, Suzuki K, Niida T, Nakajima A, Seegers LM, Vergallo R, Fracassi F, Russo M, Di Vito L, Bryniarski K, McNulty I, Lee H, Kakuta T, Nakamura S, Jang IK. Layered plaque and plaque volume in patients with acute coronary syndromes. J Thromb Thrombolysis. 2023 Apr;55(3):432-438. doi: 10.1007/s11239-023-02788-9. Epub 2023 Mar 4. PMID 36869878
- [Derived] Seegers LM, Araki M, Nakajima A, Yonetsu T, Minami Y, Ako J, Soeda T, Kurihara O, Higuma T, Kimura S, Adriaenssens T, Nef HM, Lee H, McNulty I, Sugiyama T, Kakuta T, Jang IK. Sex Differences in Culprit Plaque Characteristics Among Different Age Groups in Patients With Acute Coronary Syndromes. Circ Cardiovasc Interv. 2022 Jun;15(6):e011612. doi: 10.1161/CIRCINTERVENTIONS.121.011612. Epub 2022 Jun 2. PMID 35652353
- [Derived] Araki M, Yonetsu T, Kurihara O, Nakajima A, Lee H, Soeda T, Minami Y, Higuma T, Kimura S, Takano M, Yan BP, Adriaenssens T, Boeder NF, Nef HM, Kim CJ, McNulty I, Crea F, Kakuta T, Jang IK. Age and Phenotype of Patients With Plaque Erosion. J Am Heart Assoc. 2021 Oct 5;10(19):e020691. doi: 10.1161/JAHA.120.020691. Epub 2021 Sep 25. PMID 34569250
- [Derived] Nakajima A, Subban V, Russo M, Bryniarski KL, Kurihara O, Araki M, Minami Y, Soeda T, Yonetsu T, Crea F, Takano M, Higuma T, Kakuta T, Adriaenssens T, Boeder NF, Nef HM, Raffel OC, McNulty I, Lee H, Nakamura S, Abdullakutty J, Mathew R, Sankardas MA, Jang IK. Coronary plaque and clinical characteristics of South Asian (Indian) patients with acute coronary syndromes: An optical coherence tomography study. Int J Cardiol. 2021 Nov 15;343:171-179. doi: 10.1016/j.ijcard.2021.08.048. Epub 2021 Sep 3. PMID 34487786
- [Derived] Kurihara O, Takano M, Yamamoto E, Yonetsu T, Kakuta T, Soeda T, Yan BP, Crea F, Higuma T, Kimura S, Minami Y, Adriaenssens T, Boeder NF, Nef HM, Kim CJ, Thondapu V, Kim HO, Russo M, Sugiyama T, Fracassi F, Lee H, Mizuno K, Jang IK. Seasonal Variations in the Pathogenesis of Acute Coronary Syndromes. J Am Heart Assoc. 2020 Jul 7;9(13):e015579. doi: 10.1161/JAHA.119.015579. Epub 2020 Jul 2. PMID 32611221
- [Derived] Yamamoto E, Yonetsu T, Kakuta T, Soeda T, Saito Y, Yan BP, Kurihara O, Takano M, Niccoli G, Higuma T, Kimura S, Minami Y, Ako J, Adriaenssens T, Boeder NF, Nef HM, Fracassi F, Sugiyama T, Lee H, Crea F, Kimura T, Fujimoto JG, Fuster V, Jang IK. Clinical and Laboratory Predictors for Plaque Erosion in Patients With Acute Coronary Syndromes. J Am Heart Assoc. 2019 Nov 5;8(21):e012322. doi: 10.1161/JAHA.119.012322. Epub 2019 Oct 23. PMID 31640466
- [Derived] Sugiyama T, Yamamoto E, Fracassi F, Lee H, Yonetsu T, Kakuta T, Soeda T, Saito Y, Yan BP, Kurihara O, Takano M, Niccoli G, Crea F, Higuma T, Kimura S, Minami Y, Ako J, Adriaenssens T, Boeder NF, Nef HM, Fujimoto JG, Fuster V, Finn AV, Falk E, Jang IK. Calcified Plaques in Patients With Acute Coronary Syndromes. JACC Cardiovasc Interv. 2019 Mar 25;12(6):531-540. doi: 10.1016/j.jcin.2018.12.013. PMID 30898249